CLINICAL TRIAL: NCT02808377
Title: VAGINAL NATIVE TISSUE REPAIR AUGMENTATION WITH POST OPERATIVE PLACEMENT OF SURGICAL PELVIC ORGAN PESSARY (SPOP). A MULTICENTRE SINGLE BLINDED RANDOMISED CONTROLLED STUDY
Brief Title: Native Tissue Repair With Surgical Pelvic Organ Pessary - an RCT
Acronym: NTRSPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Ivilina Pandeva, Urogynaecology Subspecialist trainee, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A094029
Record Dates: First submitted 2016-06-07; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPOP (Active Comparator): This arm will have the soft silicone pessary inserted post operatively and it will remain in-situ for 3 weeks.
  Interventions: Other: Surgical Pelvic Organ Pessary
- Non Intervention (No Intervention): Routine post operative care

INTERVENTIONS:
Other: Surgical Pelvic Organ Pessary — In participants randomized to intervention, the SPOP will be placed at the completion of surgery, following routine placement of IDC and prior to placement of vaginal pack. The SPOP is available in 4 sizes and the surgeon will select the appropriate size so that the SPOP rests snugly without undue tension inside the hymeneal remnant. The SPOP is sutured in place with 2/0 Vicryl to prevent dislodgement at the level of the hymen.
  Arms: SPOP

SUMMARY:
This is an RCT looking at the primary outcome of composite success following anterior repair with native tissue at 6, 12, 24 months in two arms. One arm will be randomised to have a soft silicone pessary inserted into the vagina post operatively for three weeks and the other will not.

DETAILED DESCRIPTION:
Prolapse of the vagina is a common problem for women and varies from mildly bothersome to very problematic. About one in ten women in the developed world will require surgery for prolapse in their lifetime. The results of surgery are not perfect and some of women will develop prolapse again or not be satisfied with the result.

In this study a soft silicone support (SPOP) is inserted into the vagina straight after prolapse surgery. Women who have agreed to the study will be randomly chosen to have the SPOP at the time of surgery. There will be 120 patients in the study; so 60 women will have the SPOP inserted.

The investigators think that SPOP will support the vagina as it heals, improving the results of surgery. There are already some studies of the SPOP with other surgeries that show improved results. The SPOP is inserted while the patient is sleeping and is removed four weeks after surgery. It is attached with two dissolving stiches to the vagina. After four weeks is will be removed in the out patient clinic without any discomfort. It is not usually painful or uncomfortable at any time.

The actual surgery the women have will not be any different had they not been in the study. All the women in the study will have the normal assessment prior to their operation, and will fill out some questionnaires about their symptoms too. All women involved in the study will come back the clinic to be seen after six months, one year and two years from the date of the surgery. This is regardless of whether they had the SPOP or not. When the women return they will be examined and complete the questionnaires again each visit.

The results of the study will be reported and published.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic pelvic organ prolapse requiring an anterior vaginal repair at the study centre.
* Currently on the hospital waiting list for vaginal native tissue repair
* Willingness to participate
* Medically fit for surgery
* 18 years or over
* Reasonable level of English to complete questionnaires
* Patients have not been recommended surgery that involves colpocliesis, mesh, or laparoscopic approach

Exclusion Criteria:

* Asymptomatic pelvic organ prolapse
* Refusal to participate
* Medically unfit for surgery
* Under 18
* Unable to complete questionnaires due to poor level of english
* Patients has been recommended surgery that involves colpocliesis, mesh, or laparoscopic approach

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Success in anterior compartment. | 6 months post operative
  Success defined as composite of success based on objective findings and subjective patient report.
  Objective anatomic success as Anterior Prolapse no greater than Stage 1 (reference point Ba <-1cm) on validated POPQ examination. Subjective success as defined as absence of 'bulge' symptom on PDFI-20 validated questionnaire.
  Failure will be defined as leading edge of anterior vaginal wall a Stage 2 or more (reference point Ba =>-1cm), or presence of 'vaginal bulge' symptom on validated questionnaire.
Success in Anterior Compartment | 12 months post operative
  Success defined as composite of success based on objective findings and subjective patient report.
  Objective anatomic success as Anterior Prolapse no greater than Stage 1 (reference point Ba <-1cm) on validated POPQ examination. Subjective success as defined as absence of 'bulge' symptom on PDFI-20 validated questionnaire.
  Failure will be defined as leading edge of anterior vaginal wall a Stage 2 or more (reference point Ba =>-1cm), or presence of 'vaginal bulge' symptom on validated questionnaire.
Success in Anterior Compartment | 24months post operative
  Success defined as composite of success based on objective findings and subjective patient report.
  Objective anatomic success as Anterior Prolapse no greater than Stage 1 (reference point Ba <-1cm) on validated POPQ examination. Subjective success as defined as absence of 'bulge' symptom on PDFI-20 validated questionnaire.
  Failure will be defined as leading edge of anterior vaginal wall a Stage 2 or more (reference point Ba =>-1cm), or presence of 'vaginal bulge' symptom on validated questionnaire.

SECONDARY OUTCOMES:
Change in POP-Q quantitative measurements from baseline | 6 months
Change in POP-Q quantitative measurements from baseline | 12 months
Change in POP-Q quantitative measurements from baseline | 24 months
Division of vaginal band | 6months
  Any patient requiring repeat procedure for division vaginal band with in 6 months post operative.
Anatomic success of any associated posterior repair procedure | 24 months post operative
  Objective anatomic success as Posterior Prolapse no greater than Stage 1 (reference point Bp <-1cm) on validated POPQ examination.
Anatomic success of any associated posterior repair procedure | 6 months
  Objective anatomic success as Posterior Prolapse no greater than Stage 1 (reference point Bp <-1cm) on validated POPQ examination.
Anatomic success of any associated posterior repair procedure | 12 months
  Objective anatomic success as Posterior Prolapse no greater than Stage 1 (reference point Bp <-1cm) on validated POPQ examination.
Anatomic success of any associated apical repair procedure | 6 months
  Objective anatomic success as apical prolapse no greater than Stage 1 (reference point C <-1cm) on validated POPQ examination.
Anatomic success of any associated apical repair procedure | 12 months
  Objective anatomic success as apical prolapse no greater than Stage 1 (reference point C <-1cm) on validated POPQ examination.
Anatomic success of any associated apical repair procedure | 24 months
  Objective anatomic success as apical prolapse no greater than Stage 1 (reference point C <-1cm) on validated POPQ examination.
Five point Patient Global Assessment of Change (PGA-C) visual analogue scale 6 months following surgery | 6 months
Five point Patient Global Assessment of Change (PGA-C) visual analogue scale 6 months following surgery | 12 months
Five point Patient Global Assessment of Change (PGA-C) visual analogue scale 6 months following surgery | 24months
Change in PISQ-IR | 6 months
  Validated patient reported outcome - pelvic organ prolapse incontinence questionnaire IUGA revised
Change in PISQ-IR | 12 months
  Validated patient reported outcome - pelvic organ prolapse incontinence questionnaire IUGA revised
Change in PISQ-IR | 24 months
  Validated patient reported outcome - pelvic organ prolapse incontinence questionnaire IUGA revised
Change in PFDI - 20 | 24 months
  Validated patient reported outcome (pelvic floor distress inventory) -
Change in PFDI-20 | 12 months
  Validated patient reported outcome (pelvic floor distress inventory) -

OTHER OUTCOMES:
Complications of surgery as per the Clavien-Dindo classification system | Peri operative

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urogynaecology, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No